CLINICAL TRIAL: NCT05381922
Title: Rare Inherited Bleedig Disorders in Children at Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Arwa Kadry Khalaf, resident doctor at pediatric department at faculty of medicine sohag university hospital, Sohag University
Other Study IDs: Soh-Med-22-05-14
Record Dates: First submitted 2022-05-15; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Rare Inherited Bleeding Disorders in Children at Sohag University Hospital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood laboratory investigation(coagulation profile- platelet function test) — blood laboratory investigation including ( complete blood count, coagulation profile, platelet function test, level of factor decrease

SUMMARY:
The RBDs are autosomal disorders, which can be manifested in homozygotes or compound heterozygotes by a severe bleeding tendency caused by a severe deficiency or dysfunction of a clotting factor . (1) During the haemostatic response the formation of primary platelet plug limits bleeding and provides a surface for clotting factors to assemble and become activated .the initial platelet plug is stabilized by fibrin monomers ,covalently cross-linked by fXIII, forming a platelet fibrin thrombus .(2-5) Defect in platelets as well as inherited deficiencies of coagulation factors including fibrinogen ,FII,fV , FVII,FX, fXI and factor FXIII deficiencies , generally lead to lifelong bleeding disorders whose severity of bleeding symptoms is heterogeneous in platelet abnormalities but generally inversely proportional to the degree of the factor deficiency in rare bleeding disorders (RBDs). (4) the prevalence of platelet defects among the general population has not been established , whereas for RBDs it range from approximately 1in 2 million to 500,000, being higher in countries where consanguineous marriages are diffused .(6)

* As a consequence of the rarity of these deficiencies ,the type and severity of bleeding symptoms ,the underlying molecular defects and the actual management of bleeding episodes are not well established . (1) Platelet defects can alter circulating platelet numbers, function or both. These conditions are typically manifested by symptoms of excessive mucocutaneous bleeding and rapid onset, excessive bleeding following invasive surgical and dental procedures or trauma. There is considerable heterogeneity in the severity of bleeding problems associated with these defects. (7) Treatment of patients with RBDs during bleeding episodes or surgery is a challenge because of the lack of experience, paucity of data, non-availability of factor concentrates for some deficiency states and the possible occurrence of severe complications .(8) Patients who are homozygotes or compound heterozygotes for a RBD frequently present with spontaneous and or injury-related bleeding. Therapy during such episodes usually includes fresh frozen plasma or specific plasma-derived factor concentrates, which potentially carry significant risks and have adverse effects. (9,10)

ELIGIBILITY:
Inclusion Criteria:

* This study included children, aged 0-18 years, attending to pediatric department at Sohag university hospital for evaluation of bleeding symptoms, family history of a bleeding disorder and/or abnormal coagulation studies, previously diagnosed to have RBDS or recent diagnosed
* Bleeding questionnaire is done during patients' clinic visit Symptoms included in this questionnaire are epistaxis , cutaneous bleeding , minor cutaneous wound , oral cavity bleeding , hematemesis , melena and hematochezia , hematuria , tooth extraction , surgical bleeding , menorrhagia , muscle hematomas or hemoarthrosis and CNS bleeding

Exclusion Criteria:

1. Patients older than 18 years.
2. Other acquired bleeding disorder
3. common inherited bleeding disorders

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Rare inherited bleedig disorders in children at sohag university hospital
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-05-13 (Estimated); Study Completion 2023-05-13 (Estimated)

PRIMARY OUTCOMES:
prevalence of rare bleeding disorders in children at sohag university hospital | 1year
  assess the pattern ,clinical picture of different types of rare bleeding disorders and complication in children attending to hematological unit at sohag university hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Nurden P, Stritt S, Favier R, Nurden AT. Inherited platelet diseases with normal platelet count: phenotypes, genotypes and diagnostic strategy. Haematologica. 2021 Feb 1;106(2):337-350. doi: 10.3324/haematol.2020.248153. PMID 33147934
- [Background] Palla R, Peyvandi F, Shapiro AD. Rare bleeding disorders: diagnosis and treatment. Blood. 2015 Mar 26;125(13):2052-61. doi: 10.1182/blood-2014-08-532820. Epub 2015 Feb 23. PMID 25712993
- [Background] Acharya SS, Coughlin A, Dimichele DM; North American Rare Bleeding Disorder Study Group. Rare Bleeding Disorder Registry: deficiencies of factors II, V, VII, X, XIII, fibrinogen and dysfibrinogenemias. J Thromb Haemost. 2004 Feb;2(2):248-56. doi: 10.1111/j.1538-7836.2003.t01-1-00553.x. PMID 14995986
- [Background] Perez Botero J, Warad DM, He R, Uhl CB, Tian S, Otteson GE, Barness RL, Olson MC, Gossman SC, Charlesworth JE, Nichols WL, Pruthi RK, Chen D. Comprehensive Platelet Phenotypic Laboratory Testing and Bleeding History Scoring for Diagnosis of Suspected Hereditary Platelet Disorders: A Single-Institution Experience. Am J Clin Pathol. 2017 Jul 1;148(1):23-32. doi: 10.1093/ajcp/aqx038. PMID 28575217